CLINICAL TRIAL: NCT03061526
Title: Spectral-domain Optical Coherence Tomography Findings in Retinal Vessel Occlusion - A Pilot Study of Detecting Ischemia in OCT
Brief Title: Spectral-domain Optical Coherence Tomography Findings in Retinal Vessel Occlusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr.med. Egbert Matthé, Principal Investigator, Technische Universität Dresden
Other Study IDs: EK 417102016
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Retinal Ischemia
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: optical coherence tomography — measurement of reflectivity in different retinal layers based on optical coherence tomography findings

SUMMARY:
Retinal vessel occlusions might lead to ischemia of the inner retina, more severe so in artery occlusions. Intracellular edema may develop and decrease transparency of those layers, showing retinal edema. In spectral domain optical coherence tomography (SD-OCT) retinal reflectivity changes as a result of retinal edema. The investigators examine the reflectivity changes of different retinal layers between healthy eyes and eyes with retinal artery occlusion and ischemic or non-ischemic vein occlusions. Aim of the study is to evaluate whether those changes can be used to measure the level of ischemia in the inner retina.

DETAILED DESCRIPTION:
Several studies tried to classify retinal ischemia due to retinal artery or vein occlusion into different grades. In some cases prognosis is dependent on grade of severity, especially in cases of retinal vein occlusion. State of the art to Diagnose the severity of retinal ischemia is lfuorescein angiography. However, this technique is invasive and might cause Problems like anaphylactic shock. Optical coherence tomography is a non-invasive technique, but up to now there is no standardized method to quantify the grade of severity of retinal ischemia in such conditions like retinal vessel occlusion. The study hope to find criteria by which such a classification can be constructed.

ELIGIBILITY:
Inclusion Criteria:

* acute Retinal vessel occlusion on one eye
* healthy contralateral eye
* examined with spectral Domain optical coherence tomography

Exclusion Criteria:

* retinal occlusion older than 1 week
* OCT Image not obtainable/missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chart Review of patients treated b/o retinal vessel occlusion, who were examined with optical coherence tomography
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
reflectivity | December 2017
  optical density of different retinal layers

CONTACTS AND LOCATIONS:
Overall Officials: Egbert Matthé, MD, Principal Investigator — Technical University Dresden
Locations (1):
- University Eye Hospital, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matthe E, Wittig D, Kuhn M, Eulitz P, Schoen K, Sandner D, Furashova O. Manual measurement of SD-OCT images of hyperreflective retinal layers in acute retinal vessel occlusion is reliable, repeatable and reproducible. Sci Rep. 2025 Oct 3;15(1):34471. doi: 10.1038/s41598-025-20086-7. PMID 41044164